CLINICAL TRIAL: NCT03511560
Title: To Understand the Impact of Immunosuppression Using Once-per-day Envarsus XR on the Effect of Total Tacrolimus Dose/Trough Level Ratio on Renal Function (eGFR) in Kidney Transplantation
Brief Title: Envarsus on the Effect of Total Tacrolimus Dose/Trough Level Ratio on Renal Function (eGFR) in Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAR6805
Record Dates: First submitted 2018-01-29; First posted 2018-04-30 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Renal Transplant Rejection; Kidney Transplant Failure and Rejection
Keywords: Envarsus XR; Tacrolimus; Kidney Transplantation
MeSH Terms: conditions — Rejection, Psychology | interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, open-label trial examining once versus twice daily tacrolimus dosing regimen using two preparations, Envarsus vs Prograf
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus, Immediate release (Active Comparator): Tacrolimus (immediate-release) will be administered twice daily per clinical judgment of supervising physician (dosing and monitoring in accordance with center protocol) to a minimum whole blood tacrolimus concentration of at least 8 ng/mL.
  Interventions: Drug: Tacrolimus
- Envarsus XR (Experimental): Envarsus XR (Tacrolimus Extended Release Oral Tablet) will be administered once daily at initial weight-based dose of 0.12 mg/kg. Dosing and monitoring thereafter predicated on clinical judgment to a minimum whole blood tacrolimus concentration of at least 8 ng/mL. When possible, patients will receive their daily dose of Envarsus using the fewest number of pills possible.
  Interventions: Drug: Tacrolimus Extended Release Oral Tablet

INTERVENTIONS:
Drug: Tacrolimus Extended Release Oral Tablet — Tacrolimus, extended-release, oral (Envarsus); 0.75 mg, 1 mg, 4 mg tablets will be administered once daily at initial weight-based dose of 0.12 mg/kg.
  Other Names: Envarsus XR
  Arms: Envarsus XR
Drug: Tacrolimus — Tacrolimus immediate-release, oral; 0.5 mg, 1 mg, 5 mg capsules will be administered twice daily per clinical judgment of supervising physician
  Other Names: Prograf
  Arms: Tacrolimus, Immediate release

SUMMARY:
This is a one year, prospective, randomized, open-label trial examining once versus twice daily tacrolimus dosing regimen using two preparations, extended-release Tacrolimus (Envarsus XR) versus twice daily Tacrolimus (Prograf). It will examine kidney function between the two groups using estimated glomerular filtration rate (eGFR) and also examine one-year kidney outcomes, including graft loss and patient death. Patients will be followed for up to 1 year during the open-label study period.

DETAILED DESCRIPTION:
Despite lower rates of acute rejection and short-term improvements in patient and graft survival, the rate of late allograft loss following kidney transplantation has remained unchanged. Achievement of therapeutic, minimally toxic, tacrolimus concentrations early (within 30 days), after transplantation, is known to be important since achieving it has been associated with a lowered risk of acute rejection. The investigators hypothesize that using extended release tacrolimus (Envarsus XR, Veloxis), will provide more stable, more effective, and less toxic levels of tacrolimus in renal allograft recipients. Therefore, the investigators propose to analyze the impact of the blood concentration normalized by the dose (C/D ratio) on kidney function after renal transplantation in experimental group that will be treated with Envarsus XR and the standard of care (SOC) group treated with twice a day tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant patient ≥ 18 years and ≤ 80 years old
2. Institutional Review Board (IRB) approved written Informed Consent and privacy language must be obtained from the subject or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
3. Recipient of a de novo kidney from a living or deceased donor.

   a. If deceased donor, a Kidney Donor Profile Index (KDPI) ≤ 85% are eligible for enrollment.
4. Willingness to comply with study protocol.
5. Previous kidney transplants will be permitted. Patients who are receiving a secondary transplant and who previously received Envarsus or who are currently on Envarsus as a component of maintenance immunosuppression and re-listed for transplant will be eligible to enroll in this study and will be randomized at the time of transplant to either cohort.
6. Subject agrees not to participate in another study while on treatment.
7. Female subject must be either:

   1. Of non-child-bearing potential,

      * Post-menopausal (defined as at least 1 year without any menses) prior to screening, or
      * Documented surgically sterile or status post-hysterectomy
   2. Or, if of childbearing potential,

      * Agree not to try to become pregnant during the study and for 90 days after the final study drug administration
      * And have a negative serum or urine pregnancy test within 7 days prior to transplant procedure
      * And, if heterosexually active, agree to consistently use two forms of highly effective birth control (at least one of which must be a barrier method) which includes consistent and correct usage of established oral contraception, established intrauterine device or intrauterine system , or barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, starting at screening and throughout the study period and for 90 days after the final study drug administration.

Exclusion Criteria:

1. Patient is known to have a positive test for latent tuberculosis (TB) and has not previously received adequate anti-microbial therapy or would require TB prophylaxis after transplant.
2. Uncontrolled concomitant infection or any unstable medical condition that could interfere with study objectives.
3. Significant liver disease, defined as having, during the past 28 days, consistently elevated aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and/or alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SPGT)) levels greater than 3 times the upper value of the normal range of the investigational site.
4. Patient who will be maintained on a non-tacrolimus-based maintenance immunosuppressive regimen following his/her transplant procedure.
5. Patient currently taking, having taken within 30 days, or who will be maintained on an mechanistic target of rapamycin (mTOR) inhibitor following his/her transplant procedure.
6. Use of an investigational study drug in the 30 days prior to the transplant procedure.
7. Contraindication or hypersensitivity to drugs or any of their components that constitute the immunosuppression regimen.
8. Known infection or seropositivity for HIV (HBsAg and Hepatitis C (HCV) positivity with negative viral load permitted).
9. Focal segmental glomerulosclerosis.
10. Subject has a current malignancy or history of malignancy (within the past 2 years), except non-metastatic basal or squamous cell carcinoma of the skin or carcinoma-in- situ of the cervix that has been successfully treated.
11. Recipient of multi-organ kidney transplants.
12. Recipient of an en bloc, adult or pediatric deceased donor kidney
13. Any condition which, in the investigator's opinion, makes the subject unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2021-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hardy, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tacrolimus, Immediate Release | Envarsus XR
Started | 25 | 25
Completed | 24 | 21
Not Completed | 1 | 4
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Transplant cancelled | 0 | 1
Not completed — Patient switched to another drug | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus, Immediate Release | Envarsus XR | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Continuous [Mean (Full Range); unit: years] | 53 [22 to 75] | 50 [20 to 75] | 52 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Total # with Diabetes [Count of Participants; unit: Participants] | 9 | 6 | 15
Total # with History of Prior Transplantation(s) [Count of Participants; unit: Participants] | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean C/D Ratio
Description: Tacrolimus metabolism was determined for all dates of tacrolimus blood trough concentration collection after renal transplantation by dividing the tacrolimus blood trough concentration (C) by the corresponding total daily tacrolimus dose (D).
  C/D ratio (ng/mL*1/mg) = blood tacrolimus trough level (ng/mL)/total daily tacrolimus dose (mg).
Time Frame: Every Month for up to 1 year
Measure: Mean (Standard Deviation); unit: ng/mL*1/mg
Arm/Group | Tacrolimus, Immediate Release | Envarsus XR
Number analyzed (Participants) | 24 | 21
ng/mL*1/mg
  Month 1 | 1.68 (1.09) | 1.47 (.98)
  Month 2 | 1.86 (.93) | 1.85 (1.07)
  Month 3 | 2.00 (1.17) | 1.95 (1.17)
  Month 6 | 1.92 (1.07) | 2.86 (2.13)
  Month 9 | 2.05 (0.91) | 2.77 (2.33)
  Month 12 | 1.92 (1.72) | 1.97 (1.6)

2. Secondary Outcome: Mean Serum Creatinine Level
Description: Serum creatinine levels were measured to assess kidney function following transplantation
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus, Immediate Release | Envarsus XR
Number analyzed (Participants) | 24 | 21
mg/dL | 1.43 (0.79) | 1.48 (0.46)

3. Secondary Outcome: Patient Survival Rate
Description: Patient survival is any subject that is known to be alive at the study conclusion.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus, Immediate Release | Envarsus XR
Number analyzed (Participants) | 24 | 21
Participants | 24 | 21

4. Secondary Outcome: Graft Survival Rate
Description: Graft survival is defined as any subject that does not fit the following definition of graft loss: subject death, re-transplantation, transplant nephrectomy, or return to dialysis for a period of ≥6 weeks by study end.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus, Immediate Release | Envarsus XR
Number analyzed (Participants) | 24 | 21
Participants | 24 | 21

5. Secondary Outcome: Number of Rejection Episodes
Description: For study purposes, diagnoses of rejection require biopsy confirmation.
Time Frame: 12 months
Measure: Number; unit: episodes
Arm/Group | Tacrolimus, Immediate Release | Envarsus XR
Number analyzed (Participants) | 24 | 21
episodes
  C4D+ antibody-mediated biopsy proven rejection | 2 | 1
  Borderline acute cellular rejection, possible antibody-mediated rejection | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year from transplantation
Arm/Group | Tacrolimus, Immediate Release | Envarsus XR
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 8/24 | 6/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus, Immediate Release (N=24) | Envarsus XR (N=21)
BK Viremia (Infections and infestations) | 6 (6) | 4 (4)
Cytomegalovirus (Infections and infestations) | 1 (1) | 1 (1)
Epstein-Barr Virus (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT03511560/Prot_SAP_000.pdf